CLINICAL TRIAL: NCT02114840
Title: Preservation vs (Repair or Not Repair) Pronator Quadratus in the Volar Plating of Distal Radial Fracture. Randomized Controlled Clinical Trial
Brief Title: Pronator Quadratus Preservation Following Volar Plate Fixation. RCT
Acronym: PROQUAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de La Frontera (Other)
Collaborators: SOCIEDAD CHILENA DE ORTOPEDIA Y TRAUMATOLOGIA (Unknown)
Responsible Party: Principal Investigator, Cristian Ricardo Correa Valencia, MD, Traumatologist/Orthopedic Surgeon, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQP-9CH
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Wrist Fracture,; Distal Radius Fracture; Pronator Quadratus; Volar Plate; Surgery
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pronator quadratus preservation (Experimental): Pronator quadratus preservation
  Interventions: Procedure: Pronator quadratus preservation after volar plate fixation in wrist fractures
- Pronator quadratus non repair (Active Comparator)
  Interventions: Procedure: Pronator quadratus nonrepair after volar plate fixation in wrist fractures
- Pronator quadratus repair after disruption (Active Comparator)
  Interventions: Procedure: Pronator quadratus repair after volar plate fixation in wrist fractures

INTERVENTIONS:
Procedure: Pronator quadratus preservation after volar plate fixation in wrist fractures — Pronator quadratus preservation after volar plate fixation in wrist fractures
  Arms: Pronator quadratus preservation
Procedure: Pronator quadratus repair after volar plate fixation in wrist fractures — Pronator quadratus repair after volar plate fixation in wrist fractures
  Arms: Pronator quadratus repair after disruption
Procedure: Pronator quadratus nonrepair after volar plate fixation in wrist fractures — Pronator quadratus nonrepair after volar plate fixation in wrist fractures
  Arms: Pronator quadratus non repair

SUMMARY:
The purpose of this study is to determine pronator quadrutus preservation have clinical impact following volar plate fixation

ELIGIBILITY:
Inclusion Criteria:

* Fractures of distal radius with instability (Aofoundation.org)
* Age between 15-75 años
* Informed consent approval for ethical comitte

Exclusion Criteria:

* Previos surgery of the hand, wrist or forearm
* Inflammatory arthropathy
* Carpal tunel syndrome
* Sensory or mixed neuropathy
* Bilater wrist fracture
* Functional deficits of ipsilateral extremity
* Functional deficits of contralateral extremity
* Complications after surgery with motor deficit
* Disease that can evolve with neuropathy during study time

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Clinical impact in dairy life | Up to 12 month
  Clinical impact in dairy life with a functional score
Pronosupination strength | Up to 12 month
  Pronosupination strength
Proprioception | Up to 12 month
  Proprioception

SECONDARY OUTCOMES:
Proprioception evolution after surgery | Up to 12 month
  Proprioception evolution after surgery
Flexor tendon rupture | Up to 12 month
Infection after surgery | Up to 12 month
  Infection after surgery
Ischaemic time surgery | Up to 12 month
  ischaemic time surgery
Pronosupination strenght evolution | Up to 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Cristian R Correa, Study Director — Universidad de La Frontera; Eduardo Guzman, Principal Investigator — Universidad de La Frontera; Pelayo Arrieta, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad de la Frontera, Hernan Henriquez Aravena Hospital, Temuco, Temuco/IX Region, Chile

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Tosti R, Ilyas AM. Prospective evaluation of pronator quadratus repair following volar plate fixation of distal radius fractures. J Hand Surg Am. 2013 Sep;38(9):1678-84. doi: 10.1016/j.jhsa.2013.06.006. Epub 2013 Aug 2. PMID 23916193
- [Result] Ries C, Maier J, Wegmann K, Zhang W, Hohendorff B, Skouras E, Muller LP, Burkhart KJ. [Anatomic relationship between the pronator quadratus and brachioradialis muscle insertion: implications for repair of the muscle after volar plate fixation of distal radius fractures]. Z Orthop Unfall. 2013 Jun;151(3):272-7. doi: 10.1055/s-0032-1328493. Epub 2013 May 21. German. PMID 23696162
- [Result] Armangil M, Bezirgan U, Basarir K, Bilen G, Demirtas M, Bilgin SS. The pronator quadratus muscle after plating of distal radius fractures: is the muscle still working? Eur J Orthop Surg Traumatol. 2014 Apr;24(3):335-9. doi: 10.1007/s00590-013-1193-2. Epub 2013 Feb 23. PMID 23435787
- [Result] Swigart CR, Badon MA, Bruegel VL, Dodds SD. Assessment of pronator quadratus repair integrity following volar plate fixation for distal radius fractures: a prospective clinical cohort study. J Hand Surg Am. 2012 Sep;37(9):1868-73. doi: 10.1016/j.jhsa.2012.06.005. Epub 2012 Jul 31. PMID 22854257
- [Result] Fallahi F, Jafari H, Jefferson G, Jennings P, Read R. Explorative study of the sensitivity and specificity of the pronator quadratus fat pad sign as a predictor of subtle wrist fractures. Skeletal Radiol. 2013 Feb;42(2):249-53. doi: 10.1007/s00256-012-1451-0. Epub 2012 Jun 9. PMID 22684408
- [Result] Hershman SH, Immerman I, Bechtel C, Lekic N, Paksima N, Egol KA. The effects of pronator quadratus repair on outcomes after volar plating of distal radius fractures. J Orthop Trauma. 2013 Mar;27(3):130-3. doi: 10.1097/BOT.0b013e3182539333. PMID 22664580
- [Result] Creteur V, Madani A, Brasseur JL. Pronator quadratus imaging. Diagn Interv Imaging. 2012 Jan;93(1):22-9. doi: 10.1016/j.diii.2011.10.006. Epub 2011 Dec 13. PMID 22277707
- [Result] Brown EN, Lifchez SD. Flexor pollicis longus tendon rupture after volar plating of a distal radius fracture: pronator quadratus plate coverage may not adequately protect tendons. Eplasty. 2011;11:e43. Epub 2011 Nov 9. PMID 22096615
- [Result] Heidari N, Clement H, Kosuge D, Grechenig W, Tesch NP, Weinberg AM. Is sparing the pronator quadratus muscle possible in volar plating of the distal radius? J Hand Surg Eur Vol. 2012 Jun;37(5):402-6. doi: 10.1177/1753193411424706. Epub 2011 Nov 8. PMID 22067296
- [Result] Zenke Y, Sakai A, Oshige T, Moritani S, Fuse Y, Maehara T, Nakamura T. Clinical results of volar locking plate for distal radius fractures: conventional versus minimally invasive plate osteosynthesis. J Orthop Trauma. 2011 Jul;25(7):425-31. doi: 10.1097/BOT.0b013e3182008c83. PMID 21464735
- [Result] Lucchina S, Fusetti C. Is early hardware removal compulsory after retention of angled drill guides in palmar locking plates? The role of pronator quadratus reconstruction. Chin J Traumatol. 2010 Apr 1;13(2):123-5. PMID 20356451
- [Result] McConkey MO, Schwab TD, Travlos A, Oxland TR, Goetz T. Quantification of pronator quadratus contribution to isometric pronation torque of the forearm. J Hand Surg Am. 2009 Nov;34(9):1612-7. doi: 10.1016/j.jhsa.2009.07.008. Epub 2009 Oct 14. PMID 19833450
- [Result] Gordon KD, Dunning CE, Johnson JA, King GJ. Influence of the pronator quadratus and supinator muscle load on DRUJ stability. J Hand Surg Am. 2003 Nov;28(6):943-50. doi: 10.1016/s0363-5023(03)00487-8. PMID 14642509
- [Result] Stuart PR. Pronator quadratus revisited. J Hand Surg Br. 1996 Dec;21(6):714-22. doi: 10.1016/s0266-7681(96)80175-6. PMID 8982912
- [Result] Sotereanos DG, McCarthy DM, Towers JD, Britton CA, Herndon JH. The pronator quadratus: a distinct forearm space? J Hand Surg Am. 1995 May;20(3):496-9. doi: 10.1016/S0363-5023(05)80116-9. PMID 7642936